CLINICAL TRIAL: NCT01616927
Title: The DIPAK 1 Study: A Randomised, Controlled Clinical Trial Assessing the Efficacy of Lanreotide to Halt Disease Progression in ADPKD
Brief Title: Study of Lanreotide to Treat Polycystic Kidney Disease
Acronym: DIPAK1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Leiden University Medical Center (Other); Erasmus Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, dr. R.T. Gansevoort, Associate Professor in Nephrology, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIPAK1; 2011-005017-37 (EudraCT Number)
Record Dates: First submitted 2012-06-06; First posted 2012-06-12 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: ADPKD; lanreotide; polycystic kidney; polycystic liver
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases; Polycystic liver disease | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard care (No Intervention): Subjects in this arm will receive standard care
- Lanreotide (Experimental)
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Lanreotide — Lanreotide will be administered once every 4 weeks as a subcutaneous injection
  Other Names: somatuline; lanreotide autogel
  Arms: Lanreotide

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is characterized by progressive cyst formation in both kidneys, in most patients leading to end stage renal disease. It is the most common hereditary renal disease with a prevalence of approximately 1 in 1,000 persons. The majority of patients also have progressive cyst formation in the liver, leading to pain, gastrointestinal discomfort and sometimes the need for liver transplantation. At present there is no proven therapeutic intervention to slow the rate of disease progression in human ADPKD. The development of renoprotective treatments that are well tolerated, is therefore of major importance.

In this respect, somatostatin analogues are promising for especially polycystic liver disease, but also for the renal phenotype. However, the studies that have been performed thus far with these agents, were underpowered and of too short duration to reach a definitive conclusion on the potential reno- and hepatoprotective efficacy of somatostatin analogues. Therefore, the present study is designed as a randomised clinical trial with sufficient duration of follow-up to investigate whether the somatostatin analogue Lanreotide slows progression of polycystic kidney and liver disease in ADPKD-patients.

To this end, 300 ADPKD patients, aged 18-60years, with an eGFR 30-60 ml/min/1.73 m2) will be randomized 1:1 to standard care or monthly subcutaneous lanreotide injections on top off standard care. These 300 subjects will go through 15 study visits in 3 years and 1 follow up visit. During these visits, questionnaires will be filled in, physical examinations will be performed, blood will be drawn and urine collected. After study completion, rate of renal function decline in lanreotide treated subjects will be compared to that of subject who received standard care.

DETAILED DESCRIPTION:
Aims:

First, to determine whether Lanreotide attenuates progression of the renal phenotype in ADPKD patients as measured by change in rate of renal function decline and change in renal volume growth.

Second, to determine whether Lanreotide modifies progression of the liver phenotype in the subset of ADPKD patients with moderate to severe polycystic liver disease as measured by change in liver volume.

Methods:

Investigator driven, randomized, multi-center, controlled clinical trial.

Study population:

300 subjects, diagnosed with ADPKD, based on the revised Ravine criteria, with advanced disease and high likelihood of rapid disease progression (eGFR between 30 and 60 ml/min/1.73 m2 and age between 18 and 60 years).

Intervention:

Patients will be randomized (1:1) into two groups. One group will receive a dose of Lanreotide 120 mg sc every 28 days for 30 months. The dose of Lanreotide will be eGFR (BSA unadjusted) dependent. Subjects that reach an eGFR <30ml/min during the study will receive Lanreotide 90 mg sc every 28 days. Down-titration will also occur in case of dose related side effects. The other group of patients will receive standard care.

Main study endpoint:

Change in renal function in Lanreotide versus not treated patients, as assessed as slope through serial eGFR measurements over time during the treatment phase of the trial, with the value obtained at month 3 as first eGFR value for slope analysis.

Main secondary outcome variables:

* to determine whether Lanreotide modifies ADPKD progression as measured by change in renal volume in the overall study population,
* to determine whether Lanreotide modifies ADPKD progression as measured by change in liver volume in the subset of ADPKD patients with moderate to severe polycystic liver disease
* to determine whether Lanreotide changes the quality of life
* to determine whether Lanreotide is well tolerated

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ADPKD, based upon the modified Ravine criteria
2. Age between 18 and 60 years.
3. eGFR (MDRD) between 30 and 60 ml/min/1.73 m2.
4. Providing informed consent.

Exclusion Criteria:

1. Patients who, in the opinion of the study investigator may present a safety risk.
2. Patients who are unlikely to adequately comply with the trial's procedures [due for instance to medical conditions likely to require an extended interruption or discontinuation, history of substance abuse or noncompliance).
3. a. Patients taking medications or having concomitant illnesses likely to confound endpoint assessments (e.g. nephrotoxic medications such as chronic NSAID, cyclosporine, lithium immunosuppressant use) b. Patients having concomitant illnesses likely to confound endpoint assessments (e.g. diabetes mellitus for which medication is needed and patients with proteinuria > 1 g /24hr).
4. Patients who underwent surgical or drainage interventions for cystic kidney disease the year before study-entry or are likely candidates for these procedures within 2 years of start of the study.
5. Patients taking other experimental (i.e.,non approved by FDA/EMA or indication of ADPKD) therapies.
6. Patients having used Lanreotide (or another somatostatin analogue) in the 3 months before study start.
7. Patients with known intolerance for Lanreotide (or another somatostatin analogue).
8. Unwillingness to comply with reproductive precautions. Women who are capable of becoming pregnant must be willing to comply with approved birth control from two-weeks prior to, and for 60 days after taking investigational product.
9. Women, who are pregnant or breastfeeding.
10. Patients, who suffer from cardiac arrhythmias, that are thought to be dangerous in combination with lanreotide administration.
11. Patients, who ever suffered from symptomatic gallstones and did not undergo cholecystectomy.
12. Patients, who have a medical history of pancreatitis.
13. Patients, who have a medical history of infected liver cysts.

In addition:

* Patients, who underwent liver cyst drainage or surgery in the year before, can enter the study, but will not be assessed for change in liver volume.
* Patients having contraindications to, or interference with MRI assessments, as dictated by local regulation, will not be allowed to undergo MR imaging. However, these patients can enter the study, but will not be assessed for change in kidney and/or liver volume.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in renal function | serial eGFR measurements from month 3 until end of treatment visit (month 30)
  Change in renal function in Lanreotide versus not treated patients, as assessed as slope through all eGFR measurements taken at study visits during the treatment phase of the trial (n=10), with the value obtained at month 3 as first eGFR value for slope analysis.

SECONDARY OUTCOMES:
change in renal volume | baseline and 3 months after end of treatment (follow-up; month 33)
  to determine whether Lanreotide modifies ADPKD progression as measured by change in renal volume in the overall study population. Renal volume is measured at baseline, after 30 months of treatment and 3 months afterwards (follow-up visit).
change in liver volume | Baseline and end of treatment (month 30)
  to determine whether Lanreotide modifies ADPKD progression as measured by change in liver volume in the subset of ADPKD patients with moderate to severe polycystic liver disease, defined as a liver volume of >2000 ml. Liver volume is measured at baseline, at month 30 and 3 months afterwards (follow-up visit))
change in quality of life | baseline-end of treatment (month 30)
  to determine whether Lanreotide changes the quality of life (using specific questionnaires). These questionnaires will be filled in at baseline, after 3 months of treatment, after 1 year, after 2 years, at end of treatment (30 months) and at follow-up (3 months after end of treatment)
tolerance | baseline-end of treatment(month 30)
  to determine whether lanreotide is safe and well tolerated. This is assessed by investigating (severe)adverse events, vital signs, performing physical examination and clinical laboratory tests.
change in renal function | baseline and 3 months after end of treatment (follow-up; month 33)
  change in renal function in Lanreotide versus not treated patients, as assessed as change in eGFR from baseline versus eGFR obtained 3 months after cessation of treatment.
Incidence of worsening renal function | from baseline
  incidence of worsening renal function defined as a 30% decrease in eGFR and/or need for renal replacement therapy computed from pre-treatment eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Ron Gansevoort, MD, PhD, Principal Investigator — University Medical Centre
Locations (4):
- Netherlands (4):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam

REFERENCES:
- [Background] Meijer E, Drenth JP, d'Agnolo H, Casteleijn NF, de Fijter JW, Gevers TJ, Kappert P, Peters DJ, Salih M, Soonawala D, Spithoven EM, Torres VE, Visser FW, Wetzels JF, Zietse R, Gansevoort RT; DIPAK Consortium. Rationale and design of the DIPAK 1 study: a randomized controlled clinical trial assessing the efficacy of lanreotide to Halt disease progression in autosomal dominant polycystic kidney disease. Am J Kidney Dis. 2014 Mar;63(3):446-55. doi: 10.1053/j.ajkd.2013.10.011. Epub 2013 Dec 15. PMID 24342522
- [Result] Lantinga MA, D'Agnolo HM, Casteleijn NF, de Fijter JW, Meijer E, Messchendorp AL, Peters DJ, Salih M, Spithoven EM, Soonawala D, Visser FW, Wetzels JF, Zietse R, Drenth JP, Gansevoort RT; DIPAK Consortium. Hepatic Cyst Infection During Use of the Somatostatin Analog Lanreotide in Autosomal Dominant Polycystic Kidney Disease: An Interim Analysis of the Randomized Open-Label Multicenter DIPAK-1 Study. Drug Saf. 2017 Feb;40(2):153-167. doi: 10.1007/s40264-016-0486-x. PMID 27995519
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Aapkes SE, de Haas RJ, Bernts LHP, Blijdorp CJ, Dekker SEI, van Gastel MDA, Meijer E, Veldman A, Drenth JPH, Gansevoort RT; DIPAK consortium. Incident Gallstones During Somatostatin Analog Treatment are Associated with Acute Biliary Complications Especially After Discontinuation. Drugs R D. 2021 Jun;21(2):179-188. doi: 10.1007/s40268-021-00342-7. Epub 2021 Mar 29. PMID 33779943
- [Derived] van Aerts RMM, Kievit W, D'Agnolo HMA, Blijdorp CJ, Casteleijn NF, Dekker SEI, de Fijter JW, van Gastel M, Gevers TJ, van de Laarschot LFM, Lantinga MA, Losekoot M, Meijer E, Messchendorp AL, Neijenhuis MK, Pena MJ, Peters DJM, Salih M, Soonawala D, Spithoven EM, Visser FW, Wetzels JF, Zietse R, Gansevoort RT, Drenth JPH; DIPAK-1 Investigators. Lanreotide Reduces Liver Growth In Patients With Autosomal Dominant Polycystic Liver and Kidney Disease. Gastroenterology. 2019 Aug;157(2):481-491.e7. doi: 10.1053/j.gastro.2019.04.018. Epub 2019 Apr 22. PMID 31022403
- [Derived] Meijer E, Visser FW, van Aerts RMM, Blijdorp CJ, Casteleijn NF, D'Agnolo HMA, Dekker SEI, Drenth JPH, de Fijter JW, van Gastel MDA, Gevers TJ, Lantinga MA, Losekoot M, Messchendorp AL, Neijenhuis MK, Pena MJ, Peters DJM, Salih M, Soonawala D, Spithoven EM, Wetzels JF, Zietse R, Gansevoort RT; DIPAK-1 Investigators. Effect of Lanreotide on Kidney Function in Patients With Autosomal Dominant Polycystic Kidney Disease: The DIPAK 1 Randomized Clinical Trial. JAMA. 2018 Nov 20;320(19):2010-2019. doi: 10.1001/jama.2018.15870. PMID 30422235
- See also: General description of the DIPAK consortium, including the DIPAK intervention study — http://www.dipak.nl